CLINICAL TRIAL: NCT00000817
Title: The Efficacy of a Standardized Acupuncture Regimen and Amitriptyline Compared With Placebo as a Treatment for Pain Caused by Peripheral Neuropathy in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CPCRA 022; 11572 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Peripheral Nervous System Disease
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Peripheral Nervous System Diseases; Amitriptyline; Pain; Acupuncture Therapy
MeSH Terms: conditions — HIV Infections; Peripheral Nervous System Diseases; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Pain | interventions — Amitriptyline; Acupuncture Points

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (1):
- 1 (Experimental): Participants will receive standardized or alternate point acupuncture treatment twice weekly for the first 6 weeks, then once weekly for the next 8 weeks, plus either oral amitriptyline or placebo daily for the entire 14 weeks.
  Interventions: Drug: Amitriptyline hydrochloride; Drug: Amitriptyline hydrochloride placebo; Procedure: Point acupuncture

INTERVENTIONS:
Drug: Amitriptyline hydrochloride — 75 mg oral tablet taken daily
Drug: Amitriptyline hydrochloride placebo — Oral placebo tablet taken daily
Procedure: Point acupuncture — Standardized or alternate acupuncture procedure

SUMMARY:
To evaluate the separate and combined efficacy of a standardized acupuncture regimen and amitriptyline on the relief of pain due to peripheral neuropathy and on the quality of life of HIV-infected patients.

Both amitriptyline, an antidepressant, and acupuncture, a Chinese medical approach that uses needles to relieve pain, have been used successfully to reduce pain in some people. It is not known how effectively these approaches relieve or reduce pain in patients with peripheral neuropathy secondary to HIV infection.

DETAILED DESCRIPTION:
Both amitriptyline, an antidepressant, and acupuncture, a Chinese medical approach that uses needles to relieve pain, have been used successfully to reduce pain in some people. It is not known how effectively these approaches relieve or reduce pain in patients with peripheral neuropathy secondary to HIV infection.

Patients are randomized to receive either standardized point acupuncture or alternate point acupuncture treatment twice weekly for the first 6 weeks, then once weekly for the next 8 weeks, plus either oral amitriptyline or placebo daily for the entire 14 weeks. Acupuncture points are located on the lower leg. Patients are evaluated at weeks 6 and 14 and are asked to keep a daily pain diary.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral therapy.
* Nonsystemic treatment of Kaposi's sarcoma.
* Maintenance with an existing regimen of analgesic medication or herbal treatment.

Concurrent Treatment: Required:

* Acupuncture.

Patients must have:

* HIV infection.
* Lower extremity peripheral neuropathy secondary to HIV infection.
* Pain for at least 2 weeks prior to study entry.
* Life expectancy of at least 6 months.

NOTE:

* Co-enrollment in other experimental protocols is permitted as long as dual participation is allowed in those protocols.

Prior Medication:

Allowed:

* Antiretroviral therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known allergy to amitriptyline (not applicable for patients at sites using an acupuncture only study design).
* EKG indicating malignant arrhythmia or cardiac conduction disturbances (not applicable for patients at sites using an acupuncture only study design).
* Prison incarceration.

Concurrent Medication:

Excluded:

* Active treatment for an acute opportunistic infection or malignancy (nonsystemic treatment of Kaposi's sarcoma is permitted).
* Other tricyclic antidepressants.
* MAO inhibitors.

Patients with the following prior conditions are excluded (not applicable for patients at sites using an acupuncture only study design):

* History of cardiac disease.
* History of seizure disorder.

Prior Medication:

Excluded within 2 weeks prior to study entry:

* MAO inhibitors.
* Tricyclic antidepressants.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 1994-11; Study Completion 1997-05 (Actual)

PRIMARY OUTCOMES:
Change in intensity of pain as measured by the daily pain diary and the global pain relief rating | At Weeks 6 and 14
Change in quality life | Throughout study
Change in neurological status | Throughout study
Permanent discontinuation of study treatment due to treatment failure | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Shlay J, Study Chair; Flaws B, Study Chair
Locations (11):
- United States (11):
  - Community Consortium of San Francisco, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - Baltimore Trials, Baltimore, Maryland
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners Research, Albuquerque, New Mexico
  - Clinical Directors Network of Region II, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Chavez C. Prickly business. The finer points of acupuncture. Posit Aware. 1995 Jan-Feb:14-5. PMID 11362204
- [Background] Shlay JC, Chaloner K, Max MB, Flaws B, Reichelderfer P, Wentworth D, Hillman S, Brizz B, Cohn DL. Acupuncture and amitriptyline for pain due to HIV-related peripheral neuropathy: a randomized controlled trial. Terry Beirn Community Programs for Clinical Research on AIDS. JAMA. 1998 Nov 11;280(18):1590-5. doi: 10.1001/jama.280.18.1590. PMID 9820261